CLINICAL TRIAL: NCT01454349
Title: A Randomized Dose-Escalation, Multicenter Safety and Efficacy Study of a Single Transrectal Intraprostatic Treatment of PRX302 for Lower Urinary Tract Symptoms (LUTS) Secondary to Benign Prostatic Hyperplasia (BPH)
Brief Title: Study of PRX302 for Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sophiris Bio Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRX302-2-06
Record Dates: First submitted 2011-09-27; First posted 2011-10-19 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia; BPH; Enlarged prostate; Lower urinary tract symptoms (LUTS)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — PRX302

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRX302 (Experimental)
  Interventions: Drug: PRX302
- Inactive substance (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRX302 — Single intraprostatic injection with an ascending dose per cohort of 0.75, 1.5, 3.0, and 6.0 µg/mL
  Arms: PRX302
Drug: Placebo — Single intraprostatic injection of matching placebo
  Arms: Inactive substance

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of a single treatment of PRX302 for the treatment of Benign Prostatic Hyperplasia (BPH) as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Lower Urinary Tract Symptoms (LUTS) attributable to BPH for ≥6 months
* Written informed consent prior to enrollment in the study
* IPSS ≥12
* Prostate volume of 30 - 100 mL as determined by TRUS
* Maximum urine flow (Qmax) of 4 - 15 mL/sec
* Refractory, intolerant or refused the use of alpha-blockers and/or 5 alpha-reductase inhibitors
* Unwilling or unable to undergo conventional surgical or available minimally invasive treatments
* Blood PSA values <10 ng/mL

Exclusion Criteria:

* Inability to void at least 125 mL of urine
* PVR volume >200 mL
* Presence of or history of certain conditions that could interfere with study results or endanger subject
* Use of certain prescribed medications that could interfere with study results

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety | Month 3
  Safety of PRX302
Tolerability | Month 3
  Tolerability of PRX302

SECONDARY OUTCOMES:
Efficacy | Month 3
  Efficacy of PRX302 assessed by International Prostate Symptom Score (IPSS)
Efficacy | Month 12
  Efficacy of PRX302 assessed by Qmax
Pharmacokinetics | Day 1
  Pharmacokinetics (PK) measurements of PRX302
Safety | Month 12
  Safety of PRX302
Tolerability | Month 12
  Tolerability of PRX302
Efficacy | Month 3
  Efficacy of PRX302 assessed by uroflowmetry (Qmax)
Efficacy | Month 12
  Efficacy of PRX302 assessed by IPSS

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Yocum, MD, Study Director — Sophiris Bio Corp
Locations (15):
- United States (15):
  - South Orange County Medical Research Center, Laguna Hills, California
  - Atlantic Urology Medical Group, Long Beach, California
  - California Professional Research, Newport Beach, California
  - University of Colorado Denver, Aurora, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Northwestern University, Chicago, Illinois
  - The Iowa Clinic, West Des Moines, Iowa
  - Accumed Research Associates, Garden City, New York
  - University Urology Associates, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - TriState Urological Services, Cincinnatti, Ohio
  - Urologic Consultants of SE Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Research Across America, Carrollton, Texas
  - UT Southwestern Medical Center, Dallas, Texas